CLINICAL TRIAL: NCT05474924
Title: The Role of Budesonide Intrapolyp Injection in Chronic Rhinosinusitis With Nasal Polyps. A Randomized Clinical Trial.
Brief Title: The Role of Budesonide Intrapolyp Injection in CRSwNP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ibrahim M. Gehad, ENT Specialist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50-7-7
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: CRS; Polyp, Nasal
Keywords: budesonide; CRSwNP; chronic Rhinosinusitis; Nasal polyps; Intrapolyp injection
MeSH Terms: conditions — Nasal Polyps | interventions — Budesonide; Prednisolone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Budesonide Intrapolyp injection (Experimental): patients are to receive Endoscopic Intrapolyp steroid injection weekly for 5 weeks, using the following technique, where 2 nasal packs soaked in xylometazoline hydrochloride 0.1% " Otrivin adult nasal drops" applied one pack in each nostril for 5 minutes before injection, then using the 0° nasal endoscopy patients receive intrapolyp budesonide injection by 0.5 mg/ml budesonide respules "commercially available as Pulmicort ampules" 1 ml for each nostril using 1 cc 28 gauge needle sterile syringe, where injections carefully distributed amongst visible polyps avoiding visible vessels, No local anesthesia will be used before injections, patients come back to the clinic weekly to complete a series of 5 injections.
  Interventions: Drug: Budesonide intrapolyp injection
- budesonide wash (Active Comparator): patients will be instructed to perform budesonide nasal wash, through a 250 ml squeeze bottle filled with saline, 0.5 mg/ml budesonide "Pulmicort ampule" added to the solution and half the amount used for each nostril, patients gurgle with antiseptic solution to minimize the risk of oral candidiasis, patients carry out the wash twice daily for one month duration
  Interventions: Drug: Budesonide nasal wash
- Oral steroid (Active Comparator): patients receive oral prednisolone 1 mg/kg/d tapering it by 5 mg/day for 2 weeks, patients will be prescribed omeprazole 20mg protective against gastrointestinal effects of steroid
  Interventions: Drug: Prednisolone tablets

INTERVENTIONS:
Drug: Budesonide intrapolyp injection — intrapolyp injection of budesonide in cases of nasal polyps and assessment of side effects compared to systemic steroids
  Other Names: pulmicort
  Arms: Budesonide Intrapolyp injection
Drug: Budesonide nasal wash — Budesonide Nasal wash in cases of nasal polyp 0.5 mg/2ml added to 250 ml normal saline using squeeze bottle.
  Other Names: pulmicort
  Arms: budesonide wash
Drug: Prednisolone tablets — oral prednisolone tablet dosage 1 mg/kg/d tapered daily for 2 weeks.
  Other Names: solupred
  Arms: Oral steroid

SUMMARY:
Chronic rhinosinusitis with nasal polyps is a common nasal comorbidity with a wide range of symptoms that might cause severe distress and disabilities for patients. Many patients undergo repeated courses of systemic steroids and are exposed to various adverse effects. many cases finally revert to surgery. Budesonide was safely used as a nasal wash in cases of nasal polyps, our aim to determine If intrapolyp injection is a better method for delivering budesonide.

DETAILED DESCRIPTION:
Chronic Rhinosinusitis with nasal polyps can be a severely debilitating disease, it's classically treated with steroids, and different methods of steroid delivery have been used for years. patients usually receive repeated courses of systemic steroids and experience many side effects. there have been trials of intrapolyp injection of steroids, especially triamcinolone acetate. these trials concluded that it's a safe intervention. Budesonide has been used as a nasal wash frequently in cases of nasal polyps, it also has been used safely as an intratympanic injection for cases of sudden hearing loss.. it's used as a systemic steroid in cases of inflammatory bowel diseases.

The aim of our study is to test whether polyp injection is a more effective method of budesonide delivery and less dependent on subjective compliance rather than irrigation, and If it has comparable results with oral systemic steroids on polyps

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 2 CRSwNP -indicated by elevated serum IgE & high absolute Eosinophilia- with nasal polyps whose
* ages between 18 and 60 years old
* who don't have any contraindications of systemic steroids such as glaucoma, peptic ulcer, acute psychosis, chronic infections, severe osteoporosis, severe hypertension, uncontrolled diabetes mellitus, history of thromboembolic events

Exclusion Criteria:

* cystic fibrosis
* ciliary dyskinesia,
* antrochoanal polyp
* fungal sinusitis,
* unilateral nasal polyps, a
* patients who took systemic steroids in the last 6 months before our study were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 Score | 3 months
  as a subjective method to assess the patients' quality of life "QOL" and the severity of the disease prior to treatment and after.
  All patients will fill the 22 item questionnaire where the severity of each symptom was determined by 5 point scale where 0 "no problem", 1" very mild problem", 2 "mild or slight problem", 3 "moderate problem", 4 "severe problem", 5" Problem as bad as it can be" Where the sum of each individual item score provides the SNOT-22 score

SECONDARY OUTCOMES:
Lund Mackay score | 3 months
  Mackay CT score as a tool for radiological evaluation of patients with nasal polyps where each sinus is solitary assigned a score from 0 to 2 where 0 = is no opacity , 1 = partial opacity, 2 = complete opacity, where the Osteomeatal complex is given only 0 or 2, each side is evaluated on its own and the sum of all sinus is calculated. A combined score of 24 is the maximum.

OTHER OUTCOMES:
total nasal polyp score | 3 months
  the total nasal polyp score "TNPS" will be used were polyp size evaluated through endoscopy and given a score from 0 to 3 where 0 = no visible polyps, 1= mild polyposis " polyps not reaching the upper edge of the inferior turbinate", 2= moderate polyposis " polyps reaching beyond the upper edge but not the lower edge of inferior turbinate", 3= severe polyposis " polyps reaching below the lower edge of the inferior turbinate or reaching the floor of the nose" TNPS calculated as the sum of the score on each side
Total Serum IgE | 3 months
  Serum IgE of patients in all groups will be measured before the start, after course completion and after 3 months of receiving treatment
the morning plasma cortisol level | 1 month
Absolute Eosinophilic count | 3 months
  absolute eosinophilic count of patients in all groups will be measured before the start, after course completion and after 3 months of receiving treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University hospital, Kafrelsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang TW, Chung JH, Cho SH, Lee SH, Kim KR, Jeong JH. The Effectiveness of Budesonide Nasal Irrigation After Endoscopic Sinus Surgery in Chronic Rhinosinusitis With Asthma. Clin Exp Otorhinolaryngol. 2017 Mar;10(1):91-96. doi: 10.21053/ceo.2016.00220. Epub 2016 Jul 21. PMID 27440128
- [Background] Kiris M, Muderris T, Yalciner G, Bercin S, Sevil E, Gul F. Intrapolyp steroid injection for nasal polyposis: Randomized trial of safety and efficacy. Laryngoscope. 2016 Aug;126(8):1730-5. doi: 10.1002/lary.25945. Epub 2016 Mar 24. PMID 27011266
- [Result] Hansen MB, Alanin MC. Injection of Steroid in Nasal Polyps: A Systematic Review. Am J Rhinol Allergy. 2020 Nov;34(6):838-845. doi: 10.1177/1945892420936198. Epub 2020 Jun 24. PMID 32579018